CLINICAL TRIAL: NCT01311297
Title: Clinical Monitoring of Endothelial Dysfunction for Pregnant Women and in the Perioperative Course - a Pilot Study
Brief Title: Clinical Monitoring of Endothelial Dysfunction for Pregnant Women and in the Perioperative Course
Status: Terminated | Type: Observational
Sponsor: Claudia Spies (Other)
Responsible Party: Sponsor-Investigator, Claudia Spies, Prof. , MD Director of the Department of Anaesthesiology and Intensive Care Medicine CVK/CCM, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Other Study IDs: POPEYE
Record Dates: First submitted 2011-03-08; First posted 2011-03-09 (Estimated); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Endothelial Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Perioperative ovarian cancer patients
- Pregnant patients
- Female healthy volunteers

SUMMARY:
A single- center prospective observational study. This study evaluates different aspects of endothelial function. It investigates the endothelial leakage with the venous occlusion plethysmography and the flow-mediated vasodilatation by ischaemia reperfusion testing.

ELIGIBILITY:
Inclusion Criteria:

* Offered patient information and written informed consent
* Female patients aged greater than or equal to 18 years:

  1. for reduction of a primary ovarian tumour or recidive of an ovarian tumour
  2. pregnant patients with:

     * clinical normal pregnancy
     * pregnancy with weight gain of more than 10 kg
     * pregnancy and gestosis
  3. healthy volunteers

Exclusion Criteria:

* Persons without the capacity to consent
* Unability of German language use
* Lacking willingness to save and hand out data within the study
* Accommodation in an institution due to an official or judicial order
* (Unclear) history of alcohol or substances disabuse
* Coworker of the Charité
* Advanced disease of the oesophagus or upper respiratory tract
* Operation in the area of the oesophagus or nasopharynx within the last two months
* Neurological or psychiatric disease
* CHF (congestive heart failure) according to (New York Heart Association) classification - NYHA class IV at the beginning of hospital stay
* American Society of Anaesthesiologists (ASA) classification greater than IV
* Renal insufficiency (dependency of haemodialysis)
* Pulmonal oedema in thorax x-ray
* History of intracranial hemorrhage within one year of participation in the study
* Conditions following venous thrombosis within the last three years before study inclusion
* Inflammatory or reflective disease of blood vessels (Raynaud-Syndrome, Vasculitis)
* Inherent connective tissue disease(e.g. Marfan Syndrome)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female patients being treated in the Department of Gynecology and Obstetrics, Campus Virchow Klinikum, Charité - Universitaetsmedizin Berlin
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2011-03-29 (Actual); Primary Completion 2012-09-29 (Actual); Study Completion 2012-09-29 (Actual)

PRIMARY OUTCOMES:
Filtration coefficient | perioperatively up to the fifth postoperative day in patients undergoing surgery
  Endothelial parameter from the examination with venous occlusion plethysmography.
Filtration coefficient | up to one hour single measurement in pregnant woman
  Endothelial parameter from the examination with venous occlusion plethysmography.

SECONDARY OUTCOMES:
All patients: Hemodynamic parameters | perioperatively up to the fifth postoperative day in patients undergoing surgery
All patients: Markers of endothelial dysfunction (ICAM-1, E-Selectin, vWF) | perioperatively up to the fifth postoperative day in patients undergoing surgery
All patients: Endothelial flow-mediated vasodilatation | perioperatively up to the fifth postoperative day in patients undergoing surgery
Perioperative patients: Blood loss | perioperatively up to the fifth postoperative day in patients undergoing surgery
Perioperative patients: Parameter of monitored sedation (BIS - Monitoring) | during the operation
Perioperative patients: Incidence and impact of organ dysfunctions | perioperatively up to the fifth postoperative day in patients undergoing surgery
Perioperative patients: Pain | perioperatively up to the fifth postoperative day in patients undergoing surgery
  Patient self-assessed postoperative pain levels during rest using an unmarked zero to one hundred mm visual analog scale (VAS)
Perioperative patients: Body weight | perioperatively up to the fifth postoperative day in patients undergoing surgery
Perioperative patients: Satisfaction of the patients, surgeon and anesthesiologist | on the day of surgery
Perioperative patients: Duration until clinical discharge criteria were satisfied | perioperatively up to the fifth postoperative day in patients undergoing surgery
  Postanesthesia Discharge Scoring System (PADS) for Determining Home-Readiness
Perioperative patients: Intensive care unit average length of stay; hospital average length of stay | perioperatively up to the fifth postoperative day in patients undergoing surgery
Perioperative patients: Quality of life | perioperatively up to hospital discharge in patients undergoing surgery, an expexcted average of two weeks
  Descriptive system of health-related quality of life states consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which can take one of three responses. The responses record three levels of severity (no problems/some or moderate problems/extreme problems) within a particular EQ-5D dimension.
Pregnant patients: History data of the pregnancy, parameter of Gestosis | up to one hour single measurement in pregnant woman
  Gestosis: toxemia of pregnancy
All patients: Immunological Markers | perioperatively up to the fifth postoperative day in patients undergoing surgery
  Differences in selected immunologic parameters among others IL-6, IL-10

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, Campus Virchow Klinikum, Charité - Universitaetsmedizin, Berlin, Germany

REFERENCES:
- [Derived] Feldheiser A, Dathe JJ, Heinig S, Peitzner K, Kaufner L, Hunsicker O, von Haefen C, Sehouli J, Spies C. Perioperative micro-arterial function and extravasation in cytoreductive ovarian cancer surgery: an observational study. Intensive Care Med Exp. 2026 Jan 25;14(1):7. doi: 10.1186/s40635-025-00839-4. PMID 41580514